CLINICAL TRIAL: NCT02934178
Title: A Phase 1 Randomized, Double-Blinded, Placebo-controlled, Dose-Escalation Study to Assess the Safety, Tolerability and Immunogenicity of Live Attenuated, Oral Shigella WRSS1 Vaccine in Bangladeshi Toddlers (12 to 24 Months Old)
Brief Title: Shigella WRSS1 Vaccine Trial in Bangladesh
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-049
Record Dates: First submitted 2016-08-30; First posted 2016-10-14 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Diarrhea
Keywords: shigellosis; Enterobacteriaceae Infections; Gram-Negative Bacterial Infections; Bacterial Infections; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary; Enterobacteriaceae Infections; Gram-Negative Bacterial Infections; Bacterial Infections; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: WRSS1 3 x 10³ CFU (Experimental): Healthy toddlers receiving 3 oral doses of 3 x 10³ colony-forming units (CFU) of Shigella sonnei Strain WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Shigella sonnei Strain WRSS1 Vaccine
- Cohort 2: WRSS1 3 x 10⁴ CFU (Experimental): Healthy toddlers receiving 3 oral doses of 3 x 10⁴ CFU of Shigella sonnei Strain WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Shigella sonnei Strain WRSS1 Vaccine
- Cohort 3: WRSS1 3 x 10⁵ CFU (Experimental): Healthy toddlers receiving 3 oral doses of 3 x 10⁵ CFU of Shigella sonnei Strain WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Shigella sonnei Strain WRSS1 Vaccine
- Cohort 4: WRSS1 3 x 10⁶ CFU (Experimental): Healthy toddlers receiving 3 oral doses of 3 x 10⁶ CFU of Shigella sonnei Strain WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Shigella sonnei Strain WRSS1 Vaccine
- Cohort 1: Placebo (Placebo Comparator): Healthy toddlers receiving 3 oral doses of placebo to match 3 x 10³ WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Placebo
- Cohort 2: Placebo (Placebo Comparator): Healthy toddlers receiving 3 oral doses of placebo to match 3 x 10⁴ WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Placebo
- Cohort 3: Placebo (Placebo Comparator): Healthy toddlers receiving 3 oral doses of placebo to match 3 x 10⁵ WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Placebo
- Cohort 4: Placebo (Placebo Comparator): Healthy toddlers receiving 3 oral doses of placebo to match 3 x 10⁶ WRSS1 approximately 4 weeks apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Shigella sonnei Strain WRSS1 Vaccine — Live attenuated, oral Shigella WRSS1 vaccine
  Arms: Cohort 1: WRSS1 3 x 10³ CFU; Cohort 2: WRSS1 3 x 10⁴ CFU; Cohort 3: WRSS1 3 x 10⁵ CFU; Cohort 4: WRSS1 3 x 10⁶ CFU
Biological: Placebo — Sterile saline solution
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo

SUMMARY:
This is a research study of an experimental (investigational) live attenuated Shigella sonnei vaccine (WRSS1) to find a dose of the vaccine that is safe, tolerable, and develops an immune response. Shigella causes bloody and watery diarrhea, and infants and children living in developing countries experience the greatest consequences of this disease.

DETAILED DESCRIPTION:
The WRSS1 vaccine in will be given to healthy toddlers (12-24 months old). The first vaccination was given to toddlers in the inpatient unit and the second and third doses will be administered on an outpatient basis. A safety evaluation was performed after the first dose before enrolling subjects in subsequent cohorts to receive a higher vaccine dose.

After the study was initiated, its funder, the Bill and Melinda Gates Foundation (BMGF) made significant changes to the PATH Enteric Vaccine Initiative (EVI) portfolio and decided not to support the three higher-dose cohorts (Cohort 1, 2, and 3) planned as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children aged between 12 to 24 month of age at the time of vaccination
2. General good health as determined by the screening evaluation no greater than 30 days before admission
3. Father, mother or other legally acceptable representative (guardian) properly informed about the study, able to understand it and sign the informed consent form
4. Normal bowel habits (< 3 grade 1 or 2 stools each day; ≥ 1 grade 1 or 2 stools every 2 days)
5. Free of obvious health problems as established by medical history and clinical examination before entering into the study.
6. Parent or guardian available for the entire period of the study and reachable by study staff throughout the entire follow-up period.
7. Signed Informed Consent from the Parent or legal guardian

Exclusion Criteria:

1. Presence of a significant medical that in the opinion of the Investigator precludes participation in the study
2. Known infection with human immunodeficiency virus (HIV)
3. Presence in the serum of hepatitis A virus (HAV) or hepatitis C virus (HCV) antibody.
4. History of congenital abdominal disorders, intussusception, abdominal surgery or any other congenital disorder.
5. Participation in research involving another investigational product (defined as receipt of investigational product) 30 days before planned date of first vaccination or concurrently participating in another clinical study, at any time during the study period, in which the child has been or will be exposed to an investigational or a non-investigational product
6. Clinically significant abnormalities on physical examination
7. Clinically significant abnormalities in screening hematology, serum chemistry as determined by the PI or the PI in consultation with the Study Physician
8. History of febrile illness within 48 hours prior to vaccination
9. Known or suspected impairment of immunological function based on medical history and physical examination
10. Prior receipt of any Shigella vaccine
11. Fever at the time of immunization. Fever is defined as a temperature ≥ 37.5C (99.5F) on axillary, oral, or tympanic measurement
12. History of known shigellosis, chronic diarrhea/dysentery in the past 2 months
13. Current use of iron or zinc supplements within the past 7 days; current use of antacids (H2 blockers, omeprazol, OTC agents) or immunosuppressive drug
14. Allergy to quinolone, sulfa, and penicillin classes of antibiotics
15. Clinical evidence of active gastrointestinal illness
16. Prior receipt of a blood transfusion or blood products, including immunoglobulins
17. Presence of any significant systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would endanger the participant's health or is likely to result in non-conformance to the protocol.
18. History of any neurologic disorders or seizures.
19. Acute disease at the time of enrolment
20. Medically significant malnutrition, defined as moderate malnutrition (wt-for-age z-score between -3.0 and -2.0) and severe malnutrition (wt-for-age z-score <-3.0 or edema)
21. Any conditions which, in the opinion of the investigator, might jeopardize the safety of study participants or interfere with the evaluation of the study objectives
22. Receipt of antimicrobial drugs for any reason or a fever ≥ 38C within 7 days before vaccination
23. History of diarrhea during the 7 days before vaccination.
24. Has any household member(s) who is immunocompromised or under the age of 1 year old.
25. Culture or polymerase chain reaction (PCR) positive for any Shigella strain

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubhana Raqib, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Mirpur Field Office, Mirpur, Bangladesh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-site study conducted in Bangladesh. The study originally planned to enroll up to 64 toddlers to receive three doses of 3x10^3, 3x10^4, 3x10^5 or 3x10^6 colony-forming units (CFU) live attenuated, oral shigella WRSS1 vaccine or placebo, however enrollment was terminated after the first dose cohort was enrolled.
Groups:
- Cohort 1: WRSS1 3x10³ CFU: Healthy toddlers received 3 oral doses of 3x10³ colony-forming unit (CFU) Shigella sonnei strain WRSS1 vaccine approximately 4 weeks apart.
- Cohort 1: Placebo: Healthy toddlers received 3 oral doses of placebo to WRSS1 approximately 4 weeks apart.
Period: Received Vaccination 1
Arm/Group | Cohort 1: WRSS1 3x10³ CFU | Cohort 1: Placebo
Started | 12 | 4
Completed | 12 | 4
Not Completed | 0 | 0
Period: Received Vaccination 2
Arm/Group | Cohort 1: WRSS1 3x10³ CFU | Cohort 1: Placebo
Started | 12 | 4
Completed | 12 | 3
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: Received Vaccination 3
Arm/Group | Cohort 1: WRSS1 3x10³ CFU | Cohort 1: Placebo
Started | 12 | 3
Completed | 11 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: WRSS1: Healthy toddlers received 3 oral doses of 3x10³ CFU Shigella sonnei strain WRSS1 vaccine approximately 4 weeks apart.
- Cohort 1: Placebo: Healthy toddlers received 3 oral doses of placebo to WRSS1 vaccine approximately 4 weeks apart.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.4 (3.03) | 16.0 (1.41) | 17.1 (2.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 76.0 (4.01) | 74.0 (2.16) | 75.5 (3.68)
Weight [Mean (Standard Deviation); unit: kilograms] | 9.6 (0.92) | 9.0 (0.34) | 9.4 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Reactogenicity by Vaccination
Description: All toddlers were monitored for evidence of immediate reactions, assessed for systemic reactogenicity (fever, irritability, decreased appetite, and decreased activity) and gastrointestinal (GI) symptoms (abdominal pain, nausea, vomiting, loose stool, diarrhea, dysentery, bloating, excess flatulence, constipation) during the 72 hours following each vaccine dose.
Time Frame: 72 hours after each vaccination (Day 3, Day 31, Day 59)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 12 | 4
Participants
  Fever: Mild | 1 | 0
  Fever: Moderate | 0 | 0
  Fever: Severe | 0 | 0
  Fever: Life Threatening | 0 | 0
  Fever: None | 11 | 4
  Decreased appetite: Mild | 0 | 0
  Decreased appetite: Moderate | 0 | 0
  Decreased appetite: Severe | 0 | 0
  Decreased appetite: Life Threatening | 0 | 0
  Decreased appetite: None | 12 | 4
  Irritability: Mild | 0 | 0
  Irritability: Moderate | 0 | 0
  Irritability: Severe | 0 | 0
  Irritability: Life Threatening | 0 | 0
  Irritability: None | 12 | 4
  Decreased activity: Mild | 0 | 0
  Decreased activity: Moderate | 0 | 0
  Decreased activity: Severe | 0 | 0
  Decreased activity: Life Threatening | 0 | 0
  Decreased activity: None | 12 | 4
  Abdominal pain: Mild | 0 | 1
  Abdominal pain: Moderate | 0 | 0
  Abdominal pain: Severe | 0 | 0
  Abdominal pain: Life Threatening | 0 | 0
  Abdominal pain: None | 12 | 3
  Nausea: Mild | 0 | 0
  Nausea: Moderate | 0 | 0
  Nausea: Severe | 0 | 0
  Nausea: Life Threatening | 0 | 0
  Nausea: None | 12 | 4
  Vomiting: Mild | 0 | 0
  Vomiting: Moderate | 0 | 0
  Vomiting: Severe | 0 | 0
  Vomiting: Life Threatening | 0 | 0
  Vomiting: None | 12 | 4
  Loose stool: Mild | 5 | 0
  Loose stool: Moderate | 0 | 0
  Loose stool: Severe | 0 | 0
  Loose stool: Life Threatening | 0 | 0
  Loose stool: None | 7 | 4
  Diarrhea: Mild | 1 | 1
  Diarrhea: Moderate | 0 | 0
  Diarrhea: Severe | 0 | 0
  Diarrhea: Life Threatening | 0 | 0
  Diarrhea: None | 11 | 3
  Dysentery: Mild | 0 | 0
  Dysentery: Moderate | 0 | 0
  Dysentery: Severe | 0 | 0
  Dysentery: Life Threatening | 0 | 0
  Dysentery: None | 12 | 4
  Bloating: Mild | 0 | 0
  Bloating: Moderate | 0 | 0
  Bloating: Severe | 0 | 0
  Bloating: Life Threatening | 0 | 0
  Bloating: None | 12 | 4
  Excess flatulence: Mild | 0 | 0
  Excess flatulence: Moderate | 0 | 0
  Excess flatulence: Severe | 0 | 0
  Excess flatulence: Life Threatening | 0 | 0
  Excess flatulence: None | 12 | 4
  Constipation: Mild | 0 | 0
  Constipation: Moderate | 0 | 0
  Constipation: Severe | 0 | 0
  Constipation: Life Threatening | 0 | 0
  Constipation: None | 12 | 4

2. Primary Outcome: Number of Participants With Adverse Events Occurring Within 28 Days After Any Vaccination by Maximum Severity
Description: All toddlers were monitored for the occurrence of any adverse event (AE) or serious adverse event (SAE). Toddlers visited the clinic for safety assessments approximately one month after each vaccination.
  Grades are based on maximum severity per participant.
Time Frame: Up to 28 days after any vaccination (up to Day 84)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 12 | 4
Participants
  Any adverse events: Mild | 5 | 3
  Any adverse events: Moderate | 6 | 1
  Any adverse events: Severe | 0 | 0
  Any adverse events: Life Threatening | 0 | 0
  Any adverse events: Death | 0 | 0
  Any adverse events: Total | 11 | 4
  AEs related to study vaccine: Mild | 0 | 0
  AEs related to study vaccine: Moderate | 0 | 0
  AEs related to study vaccine: Severe | 0 | 0
  AEs related to study vaccine: Life Threatening | 0 | 0
  AEs related to study vaccine: Death | 0 | 0
  AEs related to study vaccine: Total | 0 | 0

3. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigens
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgA antibody responses to S. sonnei Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine Invaplex-specific IgA response from circulating lymphocytes. Invaplex is a mixture of purified S. sonnei lipopolysaccharide (LPS) and purified protein antigens IpaB and IpaC.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0: number analyzed (Participants) | 9 | 2
  Day 0 | 0.09 [0.05 to 0.15] | 0.07 [0.04 to 0.12]
  Day 7: number analyzed (Participants) | 6 | 1
  Day 7 | 0.07 [0.07 to 0.08] | 0.06 [0.06 to 0.06]
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35 | 0.07 [0.07 to 0.07] | 0.07 [0.05 to 0.09]
  Day 63: number analyzed (Participants) | 9 | 3
  Day 63 | 0.07 [0.07 to 0.08] | 0.07 [0.05 to 0.09]

4. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgA antibody responses to S. sonnei lipopolysaccharide (LPS) using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants from cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine LPS-specific IgA response from circulating lymphocytes.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Cohort 1: WRSS1: Healthy toddlers received 3 oral doses of 3x10³ colony-forming unit (CFU) Shigella sonnei strain WRSS1 vaccine approximately 4 weeks apart.
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0: number analyzed (Participants) | 11 | 2
  Day 0 | 0.07 [0.07 to 0.07] | 0.06 [0.05 to 0.08]
  Day 7: number analyzed (Participants) | 8 | 1
  Day 7 | 0.07 [0.06 to 0.08] | 0.07 [0.06 to 0.07]
  Day 35 | 0.07 [0.06 to 0.08] | 0.07 [0.06 to 0.07]
  Day 63 | 0.09 [0.05 to 0.19] | 0.06 [0.06 to 0.07]

5. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgG antibody responses to S. sonnei Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine Invaplex-specific IgG response from circulating lymphocytes. Invaplex is a mixture of purified S. sonnei lipopolysaccharide (LPS) and purified protein antigens IpaB and IpaC.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.10 [0.06 to 0.18] | 0.15 [0.01 to 1.94]
  Day 7 | 0.15 [0.06 to 0.34] | 0.19 [0.01 to 2.80]
  Day 35 | 0.09 [0.07 to 0.13] | 0.11 [0.04 to 0.27]
  Day 63 | 0.14 [0.06 to 0.30] | 0.12 [0.05 to 0.29]

6. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS)
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgG antibody responses to S. sonnei LPS using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine LPS-specific IgG response from circulating lymphocytes.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.07 [0.06 to 0.07] | 0.08 [0.04 to 0.15]
  Day 7 | 0.10 [0.04 to 0.23] | 0.08 [0.06 to 0.10]
  Day 35 | 0.07 [0.07 to 0.08] | 0.08 [0.04 to 0.17]
  Day 63 | 0.11 [0.05 to 0.24] | 0.08 [0.04 to 0.16]

7. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM antibody responses to S. sonnei Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine Invaplex-specific IgM response from circulating lymphocytes. Invaplex is a mixture of purified S. sonnei lipopolysaccharide (LPS) and purified protein antigens IpaB and IpaC.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.08 [0.07 to 0.10] | 0.10 [0.03 to 0.30]
  Day 7 | 0.14 [0.05 to 0.41] | 0.09 [0.08 to 0.11]
  Day 35 | 0.08 [0.07 to 0.09] | 0.08 [0.06 to 0.12]
  Day 63 | 0.12 [0.07 to 0.20] | 0.09 [0.05 to 0.15]

8. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM antibody responses to S. sonnei LPS using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days (Days 0, 7, 35, and 63) to determine LPS-specific IgM response from circulating lymphocytes.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0: number analyzed (Participants) | 10 | 3
  Day 0 | 0.07 [0.06 to 0.08] | 0.09 [0.06 to 0.14]
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 0.13 [0.04 to 0.47] | 0.08 [0.08 to 0.09]
  Day 35: number analyzed (Participants) | 9 | 3
  Day 35 | 0.08 [0.07 to 0.10] | 0.09 [0.07 to 0.10]
  Day 63: number analyzed (Participants) | 9 | 3
  Day 63 | 0.11 [0.06 to 0.23] | 0.11 [0.04 to 0.31]

9. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigens
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7: number analyzed (Participants) | 5 | 1
  Day 7 | 1.01 [0.98 to 1.04] | 0.98 [0.98 to 0.98]
  Day 35: number analyzed (Participants) | 8 | 2
  Day 35 | 0.77 [0.43 to 1.38] | 1.00 [1.00 to 1.00]
  Day 63: number analyzed (Participants) | 8 | 2
  Day 63 | 0.79 [0.43 to 1.48] | 0.96 [0.60 to 1.55]

10. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7: number analyzed (Participants) | 8 | 1
  Day 7 | 1.00 [0.95 to 1.04] | 1.10 [1.10 to 1.10]
  Day 35: number analyzed (Participants) | 11 | 2
  Day 35 | 1.03 [0.93 to 1.14] | 1.07 [0.58 to 1.95]
  Day 63: number analyzed (Participants) | 11 | 2
  Day 63 | 1.39 [0.68 to 2.80] | 1.04 [0.51 to 2.11]

11. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.45 [0.65 to 3.24] | 1.32 [1.12 to 1.55]
  Day 35 | 0.93 [0.72 to 1.20] | 0.73 [0.14 to 3.83]
  Day 63 | 1.38 [0.48 to 3.97] | 0.82 [0.06 to 11.01]

12. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS)
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.48 [0.63 to 3.44] | 1.00 [0.42 to 2.37]
  Day 35 | 1.04 [0.99 to 1.11] | 1.07 [0.99 to 1.15]
  Day 63 | 1.58 [0.70 to 3.57] | 1.04 [1.02 to 1.06]

13. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.64 [0.53 to 5.11] | 0.90 [0.32 to 2.51]
  Day 35 | 0.98 [0.83 to 1.15] | 0.78 [0.24 to 2.56]
  Day 63 | 1.39 [0.77 to 2.49] | 0.87 [0.21 to 3.66]

14. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 1.83 [0.50 to 6.70] | 0.91 [0.61 to 1.36]
  Day 35: number analyzed (Participants) | 9 | 3
  Day 35 | 1.12 [0.93 to 1.36] | 0.93 [0.63 to 1.37]
  Day 63: number analyzed (Participants) | 9 | 3
  Day 63 | 1.58 [0.75 to 3.31] | 1.18 [0.51 to 2.71]

15. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin A (IgA) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: number analyzed (Participants) | 5 | 1
  Day 7: 4-fold rise or higher | 0 | 0
  Day 7: Less than 4-fold rise | 5 | 1
  Day 35: number analyzed (Participants) | 8 | 2
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 8 | 2
  Day 63: number analyzed (Participants) | 8 | 2
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 7 | 2
  At any time: number analyzed (Participants) | 9 | 2
  At any time: 4-fold rise or higher | 0 | 0
  At any time: Less than 4-fold rise | 9 | 2

16. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 10 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

17. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 10 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

18. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin A (IgA) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: number analyzed (Participants) | 8 | 1
  Day 7: 4-fold rise or higher | 0 | 0
  Day 7: Less than 4-fold rise | 8 | 1
  Day 35: number analyzed (Participants) | 11 | 2
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 2
  Day 63: number analyzed (Participants) | 11 | 2
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 2
  At any time: number analyzed (Participants) | 11 | 2
  At any time: 4-fold rise or higher | 1 | 0
  At any time: Less than 4-fold rise | 10 | 2

19. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin G (IgG) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 10 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

20. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin M (IgM) Antibodies in Antibody Lymphocyte Supernatant (ALS): Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 9 | 3
  Day 35: number analyzed (Participants) | 9 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 9 | 3
  Day 63: number analyzed (Participants) | 9 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 8 | 3
  At any time: number analyzed (Participants) | 10 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 8 | 3

21. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Serum: Invaplex Antigens
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgA antibody response to S. sonnei Invaplex in serum/plasma samples at Days 0, 7, 35 and 63. Invaplex is a mixture of purified S. sonnei LPS and purified protein antigens IpaB and IpaC. Serotype-specific LPS from the Walter Reed Army Institute was used to coat the enzyme-linked immunosorbent assay (ELISA) plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.17 [0.05 to 0.62] | 0.12 [0.05 to 0.28]
  Day 7 | 0.17 [0.05 to 0.58] | 0.10 [0.08 to 0.12]
  Day 35 | 0.16 [0.05 to 0.49] | 0.12 [0.04 to 0.34]
  Day 63 | 0.36 [0.05 to 2.54] | 0.13 [0.06 to 0.25]

22. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgA antibody response to S. sonnei 2a LPS in serum/plasma samples at Days 0, 7, 35 and 63. Serotype-specific lipopolysaccharide (LPS) from the Walter Reed Army Institute was used to coat the ELISA plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.10 [0.08 to 0.12] | 0.10 [0.05 to 0.21]
  Day 7 | 0.11 [0.09 to 0.12] | 0.09 [0.07 to 0.12]
  Day 35 | 0.09 [0.08 to 0.11] | 0.57 [0.00 to 1380.56]
  Day 63 | 0.32 [0.05 to 2.01] | 0.54 [0.00 to 1483.02]

23. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Serum: Invaplex Antigen
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgG antibody response to S. sonnei Invaplex in serum/plasma samples at Days 0, 7, 35 and 63. Invaplex is a mixture of purified S. sonnei LPS and purified protein antigens IpaB and IpaC. Serotype-specific LPS from the Walter Reed Army Institute was used to coat the ELISA plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 66.79 [16.02 to 278.37] | 95.23 [3.46 to 2620.02]
  Day 7 | 3.76 [0.28 to 49.97] | 82.78 [15.70 to 436.37]
  Day 35 | 146.08 [81.56 to 261.61] | 119.79 [6.35 to 2260.20]
  Day 63 | 29.44 [4.61 to 188.01] | 147.73 [10.62 to 2054.85]

24. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Serum: Lipopolysaccharide (LPS)
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgG antibody response to S. sonnei 2a LPS in serum/plasma samples at Days 0, 7, 35 and 63. Serotype-specific LPS from the Walter Reed Army Institute was used to coat the ELISA plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 5.02 [0.79 to 32.02] | 1.00 [0.00 to 2664.32]
  Day 7 | 0.68 [0.12 to 3.88] | 0.16 [0.11 to 0.25]
  Day 35 | 14.97 [3.18 to 70.47] | 1.03 [0.00 to 2926.12]
  Day 63 | 4.63 [0.69 to 30.93] | 1.06 [0.00 to 2740.34]

25. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin M (IgM) Antibodies in Serum: Invaplex Antigen
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgM antibody response to S. sonnei Invaplex in serum/plasma samples at Days 0, 7, 35 and 63. Invaplex is a mixture of purified S. sonnei LPS and purified protein antigens IpaB and IpaC. Serotype-specific LPS from the Walter Reed Army Institute was used to coat the ELISA plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 119.55 [74.94 to 190.70] | 107.03 [5.10 to 2247.74]
  Day 7 | 177.34 [109.85 to 286.29] | 116.79 [12.32 to 1107.43]
  Day 35 | 188.41 [95.77 to 370.66] | 180.28 [7.23 to 4492.80]
  Day 63 | 208.53 [121.70 to 357.30] | 198.66 [12.57 to 3140.08]

26. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin M (IgM) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgM antibody response to S. sonnei 2a LPS in serum/plasma samples at Days 0, 7, 35 and 63. Serotype-specific LPS from the Walter Reed Army Institute was used to coat the ELISA plates.
Time Frame: Days 0, 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 102.80 [74.11 to 142.58] | 108.10 [5.27 to 2217.26]
  Day 7 | 146.48 [100.59 to 213.31] | 117.38 [12.07 to 1141.64]
  Day 35 | 117.25 [86.44 to 159.03] | 174.98 [7.28 to 4206.87]
  Day 63 | 179.07 [93.31 to 343.68] | 148.62 [16.32 to 1353.41]

27. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Serum: Invaplex Antigens
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 0.97 [0.82 to 1.15] | 0.84 [0.40 to 1.76]
  Day 35 | 0.95 [0.74 to 1.20] | 0.98 [0.77 to 1.23]
  Day 63 | 2.18 [0.20 to 24.36] | 1.08 [0.89 to 1.30]

28. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.05 [0.83 to 1.33] | 0.90 [0.50 to 1.60]
  Day 35 | 0.94 [0.78 to 1.14] | 5.47 [0.00 to 6647.02]
  Day 63 | 3.18 [0.52 to 19.56] | 5.19 [0.00 to 7147.44]

29. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin G (IgG) Antibodies in Serum: Invaplex Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 0.06 [0.01 to 0.67] | 0.87 [0.12 to 6.14]
  Day 35 | 2.19 [0.70 to 6.88] | 1.26 [0.59 to 2.67]
  Day 63 | 0.45 [0.04 to 4.63] | 1.55 [0.21 to 11.37]

30. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin G (IgG) Antibodies in Serum: Lipopolysaccharide (LPS)
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 0.13 [0.01 to 2.68] | 0.16 [0.00 to 428.26]
  Day 35 | 2.98 [0.78 to 11.46] | 1.03 [0.76 to 1.38]
  Day 63 | 0.93 [0.06 to 14.47] | 1.06 [0.75 to 1.51]

31. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin M (IgM) Antibodies in Serum : Invaplex Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.48 [1.00 to 2.20] | 1.09 [0.47 to 2.51]
  Day 35 | 1.58 [0.90 to 2.77] | 1.68 [1.31 to 2.17]
  Day 63 | 1.74 [1.32 to 2.30] | 1.86 [1.28 to 2.70]

32. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin M (IgM) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7 | 1.43 [1.07 to 1.89] | 1.09 [0.51 to 2.29]
  Day 35 | 1.14 [0.78 to 1.67] | 1.62 [0.98 to 2.67]
  Day 63 | 1.74 [1.09 to 2.78] | 1.37 [0.55 to 3.46]

33. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin A (IgA) Antibodies in Serum From Baseline: Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 0 | 0
  Day 7: Less than 4-fold rise | 11 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 2 | 0
  Day 63: Less than 4-fold rise | 9 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

34. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin G (IgG) Antibodies in Serum From Baseline: Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 10 | 3
  Day 35: 4-fold rise or higher | 2 | 0
  Day 35: Less than 4-fold rise | 9 | 3
  Day 63: 4-fold rise or higher | 2 | 0
  Day 63: Less than 4-fold rise | 9 | 3
  At any time: 4-fold rise or higher | 3 | 0
  At any time: Less than 4-fold rise | 8 | 3

35. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin M (IgM) Antibodies in Serum From Baseline: Invaplex Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 1 | 0
  Day 7: Less than 4-fold rise | 10 | 3
  Day 35: 4-fold rise or higher | 2 | 0
  Day 35: Less than 4-fold rise | 9 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

36. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin A (IgA) Antibodies in Serum From Baseline: Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 0 | 0
  Day 7: Less than 4-fold rise | 11 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 2 | 0
  Day 63: Less than 4-fold rise | 9 | 3
  At any time: 4-fold rise or higher | 2 | 0
  At any time: Less than 4-fold rise | 9 | 3

37. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin G (IgG) Antibodies in Serum From Baseline: Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 2 | 0
  Day 7: Less than 4-fold rise | 9 | 3
  Day 35: 4-fold rise or higher | 2 | 0
  Day 35: Less than 4-fold rise | 9 | 3
  Day 63: 4-fold rise or higher | 4 | 0
  Day 63: Less than 4-fold rise | 7 | 3
  At any time: 4-fold rise or higher | 4 | 0
  At any time: Less than 4-fold rise | 7 | 3

38. Secondary Outcome: Count of Participants With 4-fold Rise in Immunoglobulin M (IgM) Antibodies in Serum From Baseline: Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 35, and 63
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: 4-fold rise or higher | 0 | 0
  Day 7: Less than 4-fold rise | 11 | 3
  Day 35: 4-fold rise or higher | 0 | 0
  Day 35: Less than 4-fold rise | 11 | 3
  Day 63: 4-fold rise or higher | 1 | 0
  Day 63: Less than 4-fold rise | 10 | 3
  At any time: 4-fold rise or higher | 1 | 0
  At any time: Less than 4-fold rise | 10 | 3

39. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Stool: Invaplex Antigen
Description: The mucosal immune response to the WRSS1 was evaluated by assessing fecal IgA antibody responses to S. sonnei Invaplex in ELISA assays at Days 0, 7, 28, 35, 56, 63, and 84. Invaplex is a mixture of purified S. sonnei LPS and purified protein antigens IpaB and IpaC.
Time Frame: Days 0, 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 0.78 [0.30 to 2.04] | 0.48 [0.00 to 179.80]
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 1.74 [0.82 to 3.70] | 0.65 [0.01 to 30.02]
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28 | 1.61 [0.73 to 3.54] | 1.23 [0.02 to 89.76]
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35 | 1.59 [0.68 to 3.68] | 0.61 [0.02 to 16.33]
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56 | 1.12 [0.34 to 3.63] | 1.77 [0.01 to 478.80]
  Day 63 | 1.44 [0.50 to 4.15] | 1.48 [0.28 to 7.73]
  Day 84 | 0.95 [0.33 to 2.69] | 0.52 [0.04 to 6.39]

40. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Stool: Lipopolysaccharide (LPS) Antigen
Description: The mucosal immune response to the WRSS1 was evaluated by assessing fecal IgA antibody responses to S. sonnei LPS in ELISA assays at Days 0, 7, 28, 35, 56, 63, and 84.
Time Frame: Days 0, 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
titer
  Day 0 | 1.85 [0.59 to 5.80] | 0.80 [0.02 to 41.16]
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 3.43 [1.31 to 9.04] | 0.58 [0.02 to 21.65]
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28 | 2.99 [1.33 to 6.72] | 1.53 [0.22 to 10.50]
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35 | 3.00 [1.14 to 7.88] | 0.29 [0.01 to 6.35]
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56 | 2.08 [0.62 to 6.96] | 3.51 [0.06 to 211.20]
  Day 63 | 2.05 [0.52 to 8.04] | 1.82 [0.32 to 10.50]
  Day 84: number analyzed (Participants) | 10 | 3
  Day 84 | 1.89 [0.52 to 6.83] | 0.43 [0.01 to 18.20]

41. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Stool: Invaplex Antigens
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 1.88 [0.55 to 6.48] | 1.37 [0.02 to 111.27]
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28 | 2.27 [0.48 to 10.76] | 2.58 [0.01 to 1074.70]
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35 | 1.74 [0.56 to 5.37] | 1.28 [0.01 to 194.78]
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56 | 1.44 [0.26 to 7.99] | 14.69 [0.24 to 909.75]
  Day 63 | 1.85 [0.37 to 9.34] | 3.12 [0.00 to 2395.67]
  Day 84 | 1.25 [0.26 to 5.95] | 1.10 [0.00 to 5008.88]

42. Secondary Outcome: Geometric Mean Fold Change From Baseline in Immunoglobulin A (IgA) Antibodies in Stool: Lipopolysaccharide (LPS) Antigen
Time Frame: Baseline (Day 0, pre-vaccination) and Days 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
fold change
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 1.84 [0.45 to 7.59] | 0.72 [0.00 to 108.85]
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28 | 1.64 [0.38 to 7.00] | 1.90 [0.01 to 639.87]
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35 | 1.24 [0.30 to 5.09] | 0.36 [0.00 to 334.23]
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56 | 1.14 [0.19 to 6.72] | 9.19 [0.00 to 20438.76]
  Day 63 | 1.11 [0.22 to 5.62] | 2.27 [0.01 to 420.54]
  Day 84: number analyzed (Participants) | 10 | 3
  Day 84 | 0.95 [0.16 to 5.69] | 0.53 [0.00 to 97.74]

43. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin A (IgA) Antibodies in Stool: Invaplex Antigen
Time Frame: Days 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7: 4-fold rise or higher | 3 | 1
  Day 7: Less than 4-fold rise | 7 | 2
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28: 4-fold rise or higher | 4 | 1
  Day 28: Less than 4-fold rise | 6 | 2
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35: 4-fold rise or higher | 3 | 1
  Day 35: Less than 4-fold rise | 7 | 2
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56: 4-fold rise or higher | 4 | 2
  Day 56: Less than 4-fold rise | 7 | 0
  Day 63: 4-fold rise or higher | 4 | 2
  Day 63: Less than 4-fold rise | 7 | 1
  Day 84: number analyzed (Participants) | 10 | 3
  Day 84: 4-fold rise or higher | 3 | 2
  Day 84: Less than 4-fold rise | 7 | 1
  At any time: 4-fold rise or higher | 6 | 2
  At any time: Less than 4-fold rise | 5 | 1

44. Secondary Outcome: Count of Participants With 4-fold Rise From Baseline in Immunoglobulin A (IgA) Antibodies in Stool: Lipopolysaccharide (LPS) Antigen
Time Frame: Days 7, 28, 35, 56, 63, and 84
Population: Subjects that received the vaccination on schedule and had sufficient sample to test the antigen were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
Number analyzed (Participants) | 11 | 3
Participants
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7: 4-fold rise or higher | 4 | 1
  Day 7: Less than 4-fold rise | 6 | 2
  Day 28: number analyzed (Participants) | 10 | 3
  Day 28: 4-fold rise or higher | 5 | 1
  Day 28: Less than 4-fold rise | 5 | 2
  Day 35: number analyzed (Participants) | 10 | 3
  Day 35: 4-fold rise or higher | 2 | 1
  Day 35: Less than 4-fold rise | 8 | 2
  Day 56: number analyzed (Participants) | 11 | 2
  Day 56: 4-fold rise or higher | 3 | 1
  Day 56: Less than 4-fold rise | 8 | 1
  Day 63: 4-fold rise or higher | 3 | 1
  Day 63: Less than 4-fold rise | 8 | 2
  Day 84: number analyzed (Participants) | 10 | 3
  Day 84: 4-fold rise or higher | 4 | 0
  Day 84: Less than 4-fold rise | 6 | 3
  At any time: 4-fold rise or higher | 6 | 2
  At any time: Less than 4-fold rise | 5 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected through Day 224. Non-serious adverse events are reported through 28 days after any vaccination (up to Day 84).
Arm/Group | Cohort 1: WRSS1 | Cohort 1: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/4
Other Adverse Events (participants affected / at risk) | 11/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: WRSS1 (N=12) | Cohort 1: Placebo (N=4)
Sudden death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: WRSS1 (N=12) | Cohort 1: Placebo (N=4)
Diarrhea (Gastrointestinal disorders) | 5 | 2
Mucous stools (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Furuncle (Infections and infestations) | 2 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Typhoid fever (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 0
Varicella (Infections and infestations) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02934178/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT02934178/SAP_001.pdf